CLINICAL TRIAL: NCT05940662
Title: Cost Effectiveness of Various Implant Placement Protocols in the Esthetic Zone - a Non-randomized Controlled Trial
Brief Title: Cost Effectiveness of Various Implant Placement Protocols in the Esthetic Zone
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding difficulties
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00879
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Esthetic Zone; Single Tooth Lost; Accuracy of Dental Implants; Dimensional Changes; Patient Reported Outcome Measures; Implant Survival and Success; Cost-effectiveness; Cost-Benefit Analysis; Complications; Frequency of Treatment Protocol; Single Tooth Dental Implant
Keywords: Dental implant; Digital image processing; Bone regeneration; Clinical study; Tooth extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immediate Implant Placement (Experimental): Immediate implant placement
  1. The extraction of the failing tooth will be carried out. Subsequently, immediate implant placement and bone grafting of the intra-alveolar space by the means of a well-documented xenogeneic bone substitute will be carried out, will be conducted all in one single surgical intervention.
  2. After a healing period of at least 8 weeks, implant reopening takes place (conventional loading protocol).
  Interventions: Procedure: Immediate Implant Placement
- Early Implant Placement (Experimental): Early implant placement
  1. The extraction of the failing tooth will be carried out. Within a healing period of 4-16 weeks, the extraction socket will be completely covered by soft tissues.
  2. Implant placement and bone grafting by the means of guided bone regeneration using locally harvested autogenous bone and a well-documented xenogeneic bone substitute will be carried out.
  3. After a healing period of at least 8 weeks, implant reopening takes place (conventional loading protocol).
  Interventions: Procedure: Early Implant Placement
- Late Implant Placement (Active Comparator): Late implant placement
  1. The extraction of the failing tooth and a socket grafting procedure using a well-documented xenogeneic bone substitute will be carried out. Within a healing period of at least 16 weeks, the extraction socket will be completely covered by soft tissues and complete bone healing is anticipated.
  2. Implant placement and bone grafting by the means of guided bone regeneration using locally harvested autogenous bone and a well-documented xenogeneic bone substitute will be carried out.
  3. After a healing period of at least 8 weeks, implant reopening takes place (conventional loading protocol).
  Interventions: Procedure: Late Implant Placement

INTERVENTIONS:
Procedure: Immediate Implant Placement — The extraction of the failing tooth will be carried out. Subsequently, immediate implant placement and bone grafting of the intra-alveolar space by the means of a well-documented xenogeneic bone substitute will be carried out, will be conducted all in one single surgical intervention.
  After a healing period of at least 8 weeks, implant reopening takes place (conventional loading protocol).
  Arms: Immediate Implant Placement
Procedure: Early Implant Placement — The extraction of the failing tooth will be carried out. Within a healing period of 4-16 weeks, the extraction socket will be completely covered by soft tissues.
  Implant placement and bone grafting by the means of guided bone regeneration using locally harvested autogenous bone and a well-documented xenogeneic bone substitute will be carried out.
  After a healing period of at least 8 weeks, implant reopening takes place (conventional loading protocol).
  Arms: Early Implant Placement
Procedure: Late Implant Placement — The extraction of the failing tooth and a socket grafting procedure using a well-documented xenogeneic bone substitute will be carried out. Within a healing period of at least 16 weeks, the extraction socket will be completely covered by soft tissues and complete bone healing is anticipated.
  Implant placement and bone grafting by the means of guided bone regeneration using locally harvested autogenous bone and a well-documented xenogeneic bone substitute will be carried out.
  After a healing period of at least 8 weeks, implant reopening takes place (conventional loading protocol).
  Arms: Late Implant Placement

SUMMARY:
Loss of teeth in the anterior upper jaw significantly affects both well-being and chewing function. Nowadays, dental implants are the treatment of choice for replacing missing teeth with fixed dental prostheses and are often placed in the anterior upper jaw.

Depending on various patient-related factors, protocols for the placement of dental implants involve the following time points after tooth extraction:

1. On the same day (immediate implantation)
2. After 1-4 months (early implantation)
3. After more than 4 months (late implantation).

The different treatment protocols have been investigated over long periods. The choice of the individually suitable treatment protocol for dental implantation depends on many factors and is of utmost importance in order to achieve the best possible treatment outcomes. Selecting an inappropriate treatment protocol would otherwise result in an increased risk of failure.

After decades of research and development in dental implantology, an expert association (International Team for Implantology, ITI) published an evidence-based decision management tool in 2022. This decision management tool assists dentists in choosing the individually suitable implant treatment protocol for single-tooth replacement in the upper jaw. A structured examination of the tooth to be extracted allows to classify the situation and select the most suitable treatment protocol for the individual situation. The treatment protocols differ in terms of time and material requirements, which are associated with different costs.

There is limited data about the cost-effectiveness of these treatment protocols. The present study aims to assess how the costs of the three treatment protocols differ in relation to treatment success.

DETAILED DESCRIPTION:
Tooth loss in the visible esthetic zone of the anterior maxilla strongly impairs both patients' psychosocial well-being and masticatory function with a high demand for tooth replacement. Therefore, single tooth replacement by dental implant therapy is a very frequent indication in the esthetic zone, being corroborated with high expectations on esthetic parameters of the treatment outcomes.

Depending on local, systemic, surgical, and prosthetic factors, dental implant placement can be carried out utilizing different protocols according to the time after tooth extraction: immediate (same day, fresh extraction socket), early (1-4 months, soft tissue healing), or late (more than 4 months after tooth extraction, bone healing). Insufficient weighting of risk factors may lead to the selection of a too risky implant placement protocol, which may cause implant failures in the esthetic zone. Therefore, the appropriate selection of timepoint and corresponding surgical protocol for implant placement are of outmost importance to achieve satisfying and predictable long-term treatment outcomes in the esthetic zone.

To guide clinicians in the choice of the individually appropriate placement protocol for single tooth replacement in the esthetic zone, an evidence-based decision management tool was developed and released by the International Team for Implantology (ITI) in 2022 after decades of research and developments in dental implantology. The flowchart includes radiographic and clinical pre- and intraoperative assessments when extracting a failing tooth, to apply defined inclusion/exclusion criteria to the individual case and define the indicated implant placement protocol aiming at high implant survival and success rates.

Besides the timepoint of implant placement, the implant placement protocols involve differing amount of surgeries (immediate: 1-2, early: 3, late: 3-4), techniques for tissue augmentation including varying amount of biomaterials (immediate: socket grafting (SG), early: guided bone regeneration (GBR), late: SG and GBR) and estimated overall clinical visits (immediate: minimum 4, early: minimum 5, late: minimum 6). All these factors contribute to the operating costs of a private practice/dental clinic in implant dentistry, with the majority of costs being composed of material costs and the procedural time involved.

To date, there is a lack of data about the cost effectiveness of dental implant placement using varying implant placement protocols. Therefore, this study is designed to primarily evaluate the surgical costs in relation to the implant survival rates of implant placement procedures using various placement protocols as indicated by an evidence-based decision management tool. The secondary outcomes include the assessment of placement protocol frequency, biological/mechanical/technical complication rates and the long-term stability of regenerated tissues.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Willingness and ability to sign informed consent (Appendix Informed Consent Form) and to participate in the study
* Plaque index according to Silness and Loe of < 35%
* Presence of a single tooth (FDI positions 15 - 25) that has to be extracted
* Sufficient vertical interocclusal space for the placement of an implant crown (FDI regions 13-23: 3 mm, FDI regions 15, 14, 24, 25: 6 mm)
* Ridge height sufficient for the placement of a ≥ 8 mm-long implant
* Sufficient ridge width for the placement of a 2.9 mm diameter implant (min. 5 mm)

Exclusion Criteria:

* Any physical or mental disorder that would interfere with the ability to perform adequate oral hygiene or the capability of providing written informed consent and compliance to the protocol
* Any disorder that would interfere with wound healing or represent a contraindication for implant surgery such as, but not limited to, uncontrolled diabetes or conditions resulting in or requiring immunosuppression, radiation, chemotherapy, frequent use of antibiotics or antiresorptive medication such as bisphosphonates
* Pregnancy (pregnancy tests will be applied; see chapter 6.5)
* Intention to become pregnant between inclusion and implant loading
* Heavy smoking habit with ≥ 10 cig/d
* Allergy to titanium
* Severe bruxism or clenching habits, present oro-facial pain
* Insufficient ridge width/height for the study implant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2029-01-01 (Estimated); Primary Completion 2032-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment costs | From enrollment to the 1 year follow-up
  Overall treatment costs for implant placement using three implant placement protocols
Implant survival rates | From enrollment to the 1 year follow-up
  Subordinate/Descriptive primary outcome: implant survival rates

SECONDARY OUTCOMES:
Implant success | From enrollment to the 10 year follow-up
  Absence of persisting subjective discomfort such as pain, foreign body perception and or dysaesthesia (e. g. painful sensation), absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if observed at two or more follow-up visits after the treatment with systemic antibiotics), absence of implant mobility on manual palpation, absence of any continuous peri-implant radiolucency
Frequency of application of the various types of implant placement protocols | From enrollment to the end of treatment at 8 weeks
  The frequency of application of the various types of implant placement (immediate, early, late), when applying the inclusion-criteria of a decision management tool
Complication rates | From enrollment to the 10 year follow-up
  Biological/technical/mechanical complication rates as defined by (Salvi et al., 2009; Schwarz et al., 2018)
Esthetic outcomes | From enrollment to the 10 year follow-up
  Esthetic outcomes by evaluating standardized digital photographs using pink/white esthetic scores
Patient-centered outcomes | From enrollment to the 10 year follow-up
  Patient-centered outcomes: placement protocol-related satisfaction (visual analogue scale (VAS)-based questionnaire)
Accuracy of implant position | From enrollment to the end of treatment at 8 weeks
  Accuracy of the final implant position compared of computer-assisted implant placements compared to the virtually pre-operatively planned implant position by superimposition of intraoral scans
Soft tissue stability | From enrollment to the 10 year follow-up
  Long term stability of the soft tissue dimensions utilizing digital imaging
Hard tissue stability | From enrollment to the 10 year follow-up
  Stability of the facial bone augmentation after implant placement using digital imaging
Crestal Bone Levels | From enrollment to the 10 year follow-up
  Mesial and distal implant bone level changes using standardized and digitized peri-apical radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Raabe, Principal Investigator — Klinik für Oralchirurgie und Stomatologie, Universität Bern
Locations (1):
- Klinik für Oralchirurgie und Stomatologie, zmk Bern, Universität Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
After publication some additional non-published data can be given upon reasonable request.

REFERENCES:
- [Background] Tonetti MS, Cortellini P, Graziani F, Cairo F, Lang NP, Abundo R, Conforti GP, Marquardt S, Rasperini G, Silvestri M, Wallkamm B, Wetzel A. Immediate versus delayed implant placement after anterior single tooth extraction: the timing randomized controlled clinical trial. J Clin Periodontol. 2017 Feb;44(2):215-224. doi: 10.1111/jcpe.12666. Epub 2017 Jan 31. PMID 27978602
- [Background] Ducommun J, El Kholy K, Rahman L, Schimmel M, Chappuis V, Buser D. Analysis of trends in implant therapy at a surgical specialty clinic: Patient pool, indications, surgical procedures, and rate of early failures-A 15-year retrospective analysis. Clin Oral Implants Res. 2019 Nov;30(11):1097-1106. doi: 10.1111/clr.13523. Epub 2019 Aug 30. PMID 31400242
- [Background] Buser D, Janner SF, Wittneben JG, Bragger U, Ramseier CA, Salvi GE. 10-year survival and success rates of 511 titanium implants with a sandblasted and acid-etched surface: a retrospective study in 303 partially edentulous patients. Clin Implant Dent Relat Res. 2012 Dec;14(6):839-51. doi: 10.1111/j.1708-8208.2012.00456.x. PMID 22897683
- [Background] Buser D, Chappuis V, Kuchler U, Bornstein MM, Wittneben JG, Buser R, Cavusoglu Y, Belser UC. Long-term stability of early implant placement with contour augmentation. J Dent Res. 2013 Dec;92(12 Suppl):176S-82S. doi: 10.1177/0022034513504949. Epub 2013 Oct 24. PMID 24158332
- [Background] Buser D, Chappuis V, Belser UC, Chen S. Implant placement post extraction in esthetic single tooth sites: when immediate, when early, when late? Periodontol 2000. 2017 Feb;73(1):84-102. doi: 10.1111/prd.12170. PMID 28000278